CLINICAL TRIAL: NCT00360100
Title: A Randomized, Multicenter, Comparative Study To Assess Tolerability Of A Single Oral 60 Mg/Kg Dose Of Zmax (Pediatric Concentration) Vs. Zmax (Adult Concentration) In Pediatric Patients With Acute Otitis Media
Brief Title: Zmax Pediatric Vs Adult Concentration For The Treatment Of Acute Otitis Media
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0661170
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2011-05

CONDITIONS: Otitis Media
MeSH Terms: conditions — Otitis Media | interventions — Azithromycin

INTERVENTIONS:
Drug: Zmax

SUMMARY:
Assess tolerability of different dosing formulations (adult versus pediatric).

ELIGIBILITY:
Inclusion Criteria:

* Have clinical signs/symptoms of AOM in at least 1 ear

Exclusion Criteria:

* Known or suspected hypersensitivity, or intolerance to azithromycin or other macrolides or to any penicillin, beta-lactam antibiotic or beta lactamase inhibitor
* Previously diagnosed disease(s) of immune function
* Treatment with any systemic (intravenous, intramuscular, oral) antibiotic for any indication within 7 days prior to enrollment

Ages: 3 Months to 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2006-08; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Treatment-related vomiting on Day 1, which is based directly on the collected observed or voluntarily reported vomiting.

SECONDARY OUTCOMES:
Time-to-vomiting (in minutes) will be measured for all vomiting episodes that occur within the 60-minute observation period post-dosing on Day 1.
Frequency of the number of days of treatment-related vomiting by treatment group for subjects in the All Treated population.
Frequencies of occurrence, by day, of treatment-related vomiting.
Investigator and Sponsor assessment of clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- United States (2):
  - Pfizer Investigational Site, Bardstown, Kentucky
  - Pfizer Investigational Site, Springfield, Kentucky
- Pfizer Investigational Site, Córdoba, Córdoba Province, Argentina
- Chile (3):
  - Pfizer Investigational Site, Santiago, RM
  - Pfizer Investigational Site, Independencia, Santiago Metropolitan
  - Pfizer Investigational Site, Providencia, Santiago Metropolitan
- Pfizer Investigational Site, San José, Costa Rica
- Pfizer Investigational Site, Santo Domingo, DN, Dominican Republic
- Pfizer Investigational Site, Guatemala City, Guatemala
- Pfizer Investigational Site, Panama City, Panama

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661170&StudyName=Zmax+Pediatric+Vs+Adult+Concentration+For+The+Treatment+Of+Acute+Otitis+Media++